CLINICAL TRIAL: NCT06955988
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AST2303 Tablets (ABK3376 Tablets) in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of AST2303 Tablets (ABK3376 Tablets) in Patients With Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Allist Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALSC001AST2303
Record Dates: First submitted 2025-04-11; First posted 2025-05-02 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: EGFR L858R-C797S; Del19-C797S
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- AST2303 Tablets(ABK3376 Tablets) ，25mg (Experimental): AST2303 Tablets(ABK3376 Tablets) ，25mg
  Interventions: Drug: AST2303 Tablets(ABK3376 Tablets) ，25mg
- AST2303 Tablets(ABK3376 Tablets) ，50mg (Experimental): AST2303 Tablets(ABK3376 Tablets) ，50mg
  Interventions: Drug: AST2303 Tablets(ABK3376 Tablets) ，50mg
- AST2303 Tablets(ABK3376 Tablets) ，75mg (Experimental): AST2303 Tablets(ABK3376 Tablets) ，75mg
  Interventions: Drug: AST2303 Tablets(ABK3376 Tablets) ，75mg
- AST2303 Tablets(ABK3376 Tablets) ，100mg (Experimental): AST2303 Tablets(ABK3376 Tablets) ，100mg
  Interventions: Drug: AST2303 Tablets(ABK3376 Tablets) ，100mg
- AST2303 Tablets(ABK3376 Tablets) ，125mg (Experimental): AST2303 Tablets(ABK3376 Tablets) ，125mg
  Interventions: Drug: AST2303 Tablets(ABK3376 Tablets) ，125mg

INTERVENTIONS:
Drug: AST2303 Tablets(ABK3376 Tablets) ，25mg — Usage and dosage: 25mg, oral on an empty stomach Duration of medication: oral once a day, 21 days as a cycle
  Arms: AST2303 Tablets(ABK3376 Tablets) ，25mg
Drug: AST2303 Tablets(ABK3376 Tablets) ，50mg — Usage and dosage: 50mg, oral on an empty stomach Duration of medication: oral once a day, 21 days as a cycle
  Arms: AST2303 Tablets(ABK3376 Tablets) ，50mg
Drug: AST2303 Tablets(ABK3376 Tablets) ，75mg — Usage and dosage: 75mg, oral on an empty stomach Duration of medication: oral once a day, 21 days as a cycle
  Arms: AST2303 Tablets(ABK3376 Tablets) ，75mg
Drug: AST2303 Tablets(ABK3376 Tablets) ，100mg — Usage and dosage: 100mg, oral on an empty stomach Duration of medication: oral once a day, 21 days as a cycle
  Arms: AST2303 Tablets(ABK3376 Tablets) ，100mg
Drug: AST2303 Tablets(ABK3376 Tablets) ，125mg — Usage and dosage: 125mg, oral on an empty stomach Duration of medication: oral once a day, 21 days as a cycle
  Arms: AST2303 Tablets(ABK3376 Tablets) ，125mg

SUMMARY:
This study is a multicenter, single arm, open label, phase I clinical trial, including dose escalation (phase IA) and dose expansion (phase IB). This study aimed to evaluate the safety, tolerability, PK characteristics and preliminary antitumor activity of ast2303 tablets (abk3376 tablets) in subjects with locally advanced or metastatic non-small cell lung cancer. A safety review committee (SRC) was established in this study, which will review the safety, efficacy, pharmacokinetics and other data obtained from the study, and make decisions on key issues such as dose escalation and dose expansion.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood this test and voluntarily sign the informed consent
2. Age ≥ 18 at the time of signing the informed consent, regardless of gender
3. Patients with non-small cell lung cancer confirmed by tissue / cytology.
4. According to recist1.1 criteria, the presence of at least one target lesion without local treatment was assessed by the investigator
5. Agree to provide blood samples and / or tumor tissue samples (fresh tissue or paraffin embedded tissue) for genetic testing
6. The subject's bone marrow and organ functions are good (no blood transfusion or hematopoietic growth factor treatment within 2 weeks before the first administration)
7. The ECoG physical status score is 0 or 1
8. Expected survival time ≥ 12 weeks
9. Have normal swallowing function
10. Female subjects with fertility must have a serum pregnancy test within 7 days before the first administration, and the result is negative, and must be non lactating. For female subjects with fertility and male subjects with reproductive potential, effective contraceptive measures were taken from the signing of informed consent to 6 months after the last Administration

Exclusion Criteria:

1. Previously received antitumor therapy targeting the c797s mutation
2. Carry any other known driver gene alterations
3. Have received any systemic anti-tumor treatment (including anti-tumor drugs in clinical research stage) within 2 weeks before the first administration or within 5 half lives of the drug (whichever is longer); Or receiving anti-tumor drugs with long half-life, such as immune checkpoint inhibitors, within 4 weeks before the first administration; Or received cytotoxic drugs with significant delayed toxicity, such as mitomycin C, within 6 weeks before the first administration;
4. Have received non-specific immunomodulatory agents, traditional Chinese medicine or traditional Chinese medicine preparations with approved anti-tumor indications within 2 weeks before the first administration
5. Strong inhibitors of CYP3A, P-gp or BCRP were used within 7 days before the first administration, or strong inducers of CYP3A, P-gp or BCRP were used within 3 weeks
6. Local (non bone lesions) radiotherapy within 4 weeks before the first dose, or bone radiotherapy within 2 weeks before the first dose;
7. Other malignant tumors besides the primary tumor
8. Subjects known to have meningeal metastasis, brainstem metastasis, spinal cord metastasis and / or compression, active brain metastasis. For brain metastasis subjects who have received local treatment in the past, if they are clinically stable for at least 4 weeks before the first administration of study treatment and do not need to use glucocorticoids or anticonvulsants for at least 14 days before the first administration of study treatment, they can participate in the study
9. The tumor invades the surrounding important organs and blood vessels or has the risk of esophago tracheal fistula or esophago pleural fistula
10. The toxicity of previous anti-tumor treatment has not returned to grade ≤ 1 (NCI CTCAE version 5.0 evaluation), except for grade ≤ 2 alopecia and peripheral neuropathy
11. Presence of cardiovascular and cerebrovascular disease or cardiovascular and cerebrovascular risk factors
12. Uncontrollable systemic diseases
13. There is a history of (non infectious) interstitial lung disease (ILD) or non infectious pneumonia requiring steroid treatment; Currently have ILD or non infectious pneumonia; Suspected ILD or noninfectious pneumonia that could not be excluded by imaging examination was present at screening
14. Pulmonary complications lead to clinically serious lung damage, including but not limited to the following: A. any underlying lung disease; b. Any autoimmune, connective tissue or inflammatory disease that may involve the lungs; c. Previous unilateral pneumonectomy
15. Severe acute or chronic infection
16. Being under long-term systemic corticosteroid treatment with prednisone > 10 mg/ day or equivalent anti-inflammatory active drugs or any form of immunosuppressive treatment before the first administration. Subjects who need to use bronchodilators, inhaled or topical steroids or local steroid injections for treatment or as preventive medication for hypersensitivity reactions (such as medication before CT examination, etc.) can be included in the study
17. Subjects who had undergone major surgery within 4 weeks before the first dose or were expected to undergo major surgery during the study period
18. Bleeding symptoms with significant clinical significance or obvious bleeding tendency within 4 weeks before the first administration, such as gastrointestinal bleeding, gastric ulcer bleeding, active hemoptysis, etc
19. It is known that there are serious gastrointestinal dysfunction: such as untreated recurrent diarrhea, moderate to severe atrophic gastritis, gastrointestinal obstruction, Crohn's disease, ulcerative colitis, gastrointestinal perforation, etc
20. Known to have a history of hypersensitivity to the ingredients of the preparation used in the test
21. Pregnant or lactating women or women planning to become pregnant during the study
22. In the judgment of the investigator, the subject has other factors that may affect the results of the study or cause the forced termination of the study, such as alcohol abuse, drug abuse, suffering from other serious diseases (including mental diseases) requiring combined treatment, serious abnormal laboratory test values, family or social factors and other conditions that may affect the safety of the subject or the collection of test data, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Event, AE | Up to 2 years
  AE will be classified based on the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) of the International Conference on Harmonisation of Registration Techniques for Medicinal Products for Human Use (ICH), and graded according to CTCAE 5.0.
Serious Adverse Event (SAE) | Up to 2 years
Adverse Events of Special Concern (AESI) | Up to 2 years
Objective response rate (ORR) | Up to 2 years
  ORR is defined as the proportion of subjects confirmed as CR or PR to the total number of subjects, and the confirmation of remission is based on a follow-up evaluation conducted at least 28 days apart using the RECIST v1.1 evaluation criteria.
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the sum of the proportions of subjects whose disease is confirmed to have improved (including CR, PR) or stabilized (SD) after the start of treatment.
Duration of Relief (DOR) | Up to 2 years
  DOR is defined as the time from the first recorded CR or PR to the first recorded imaging of disease progression (evaluated according to RECIST v1.1 criteria) or death from any cause (whichever occurs first) in a subject confirmed as ORR. Subjects who did not report disease progression or death during analysis will be subject to deletion on the date of the last tumor assessment.
Progression free survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of first medication to the date of first recorded disease progression (evaluated according to RECIST v1.1 criteria) or death from any cause (whichever occurs first).
Overall survival (OS) | Up to 2 years
  OS is defined as the time from the date of initial medication to the date of death from any cause (whichever occurs first). Subjects who were not reported as deceased during the analysis, or subjects who were reported dead but had an unknown date of death (i.e. missing year, month, day, etc.), will be deleted from the last known date of survival.

SECONDARY OUTCOMES:
Peak Time (Tmax) | Up to 2 years
Peak Plasma Concentration (Cmax) | Up to 2 years
From 0 to the last measurable time point t, the area under the drug time curve (AUC0-t) | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China